CLINICAL TRIAL: NCT03944486
Title: Feasibility Study of On-Track - a Digital System for Upper Limb Rehabilitation After Stroke
Brief Title: On-Track Feasibility Study of a Rehabilitation System for Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 19SM5146
Record Dates: First submitted 2019-04-29; First posted 2019-05-09 (Actual); Results first posted 2022-03-29 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Cerebrovascular Accident
Keywords: Cerebrovascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- On-Track (Other): Stroke survivors receiving the OnTrack intervention for 12 weeks consisting of arm activity tracking and self-management coaching. Assessments are done before and after the intervention.
  Interventions: Device: Feasibility of OnTrack

INTERVENTIONS:
Device: Feasibility of OnTrack — Patients to use digital application- study assessed the feasibility of the application for patients and therapists.

SUMMARY:
Feasibility study of On-Track - a digital system for upper limb rehabilitation after stroke.

Population - stroke patients over 18 years old.

DETAILED DESCRIPTION:
TITLE Feasibility study of On Track - a digital system for upper limb rehabilitation after stroke

DESIGN & METHODS Mixed methods

Aims Assess the feasibility of 'On-Track' (a new arm rehabilitation system), for use by patients, and therapists in stroke rehabilitation services.

OUTCOME MEASURES Various. (including functional and self-reported measures)

POPULATION Stroke survivors, their family/carers, clinicians, professionals and lay people working with stroke survivors.

ELIGIBILITY Participants will be stroke survivors, relatives/carers of stroke survivors, frontline healthcare workers who treat stroke survivors, managers responsible for stroke service provision and lay people with an involvement in stroke care/delivery.

Participants will be over 18.

DURATION 1- 2 years

ELIGIBILITY:
Inclusion criteria:

* Adults (aged 18 or over).
* Stroke diagnosis less than 6 months previously (first or recurrent). Some participants will be recruited from an in-patient rehabilitation ward, hence the 6-month poststroke limit.
* Arm impairment of any type or level (including weakness-including dense hemiplegia, neglect and sensory deficits). This enables better understanding of which impairment level groups could benefit or not from using the intervention, especially considering the impact it may have on people's motivation regardless of their level of impairment.
* Ability to provide informed consent.
* Reliability to communicate (verbally or non-verbally) and understand English.
* Ability to read a predefined short message.

Exclusion criteria:

* Unstable medical condition.
* Self-reported 'severe' pain in the arm affected either at rest or during movement.
* Severe oedema in the arm affected by their stroke, judged by the consenting therapist.
* Known discharge plans to a hospital other than the recruitment site or residential care in less than 7 weeks (a small proportion of patients in in-patient rehab may be in hospital for up to 12 weeks).
* Participants who are unable to engage with the intervention for a period of more than 7 consecutive days will be reviewed in a case-by-case basis by the members of the team responsible for delivering the intervention to determine if study continuation is appropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ara Darzi, MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial Collage NHS Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taylor E, Fusari G, Darzi A, Jones F. Is a novel digital system for arm and hand rehabilitation suitable for stroke survivors? A qualitative process evaluation of OnTrack. BMJ Open. 2023 Aug 18;13(8):e062119. doi: 10.1136/bmjopen-2022-062119. PMID 37597873
- [Derived] Fusari G, Gibbs E, Hoskin L, Lawrence-Jones A, Dickens D, Fernandez Crespo R, Leis M, Crow J, Taylor E, Jones F, Darzi A. What is the feasibility and patient acceptability of a digital system for arm and hand rehabilitation after stroke? A mixed-methods, single-arm feasibility study of the 'OnTrack' intervention for hospital and home use. BMJ Open. 2022 Sep 28;12(9):e062042. doi: 10.1136/bmjopen-2022-062042. PMID 36171046
- [Derived] Fusari G, Gibbs E, Hoskin L, Dickens D, Leis M, Taylor E, Jones F, Darzi A. Protocol for a feasibility study of OnTrack: a digital system for upper limb rehabilitation after stroke. BMJ Open. 2020 Mar 23;10(3):e034936. doi: 10.1136/bmjopen-2019-034936. PMID 32205375

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: August 2019 - December 2020 Participants were identified and screened by therapists at an acute setting. Recruitment followed with participants beginning their participation at the acute setting and followed up in the community. After the start of the Covid-19 pandemic, participants were identified in the acute setting but only started participation once discharged to the community.
Groups:
- OnTrack: One arm feasibility study
  Feasibility of OnTrack: Patients to use digital application- study assessed the feasibility of the application for patients and therapists.
Period: Overall Study
Arm/Group | OnTrack
Started | 24
Completed | 12
Not Completed | 12

BASELINE CHARACTERISTICS:
Groups:
- On-Track: One arm feasibility study
  Feasibility of OnTrack: Patients to use digital application- study assessed the feasibility of the application for patients and therapists.
Arm/Group | On-Track
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] — Population: Some data was not collected before participant was withdrawn
  years
    number analyzed (Participants) | 21
    (all) | 61.133 [33.5 to 82.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 24
Patient Activation Measure (PAM) [Mean (Full Range); unit: units on a scale] — 10-item survey assessing underlying knowledge, skills and confidence integral to managing own health and healthcare.
  PAM segments individuals along an empirically derived 100-point scale (0 min - 100 max, a higher score indicates a higher level of activation). Each level provides insight into an extensive array of health-related characteristics, including attitudes, motivators, and behaviors. Population: Only measuring participants who completed the intervention.
  units on a scale
    number analyzed (Participants) | 12
    (all) | 69.7 [42.9 to 100]
Motor Activity Log (MAL) [Mean (Full Range); unit: units on a scale] — Structured interview intended to examine How Much and How Well the subject uses their more-affected arm outside of the laboratory setting. Standardized questions are asked about the amount of use of their more-affected arm (Amount Scale or AS) and the quality of their movement (How Well Scale or HW) during the functional activities. Two scales are printed on sheets of paper and are placed in front of the participant during test administration. Both scales range between 0 and 5 (half scores are possible, i.e. 0.5,1.5,2.5,3.5,4.5). Higher values represent a better outcome. Population: Only measuring participants who completed the intervention.
  units on a scale
    MAL (How much): number analyzed (Participants) | 12
    MAL (How much) | 2.0 [0.39 to 4.18]
    MAL (How well): number analyzed (Participants) | 12
    MAL (How well) | 2.26 [0.38 to 4.75]
Montreal Cognitive Assessment (MoCA) [Mean (Full Range); unit: units on a scale] — Aims to test subjects with Mild Cognitive Impairment irrespective of etiology. Covers most cognitive domains and is available in 3 versions to decrease possible learning effects when the MoCA is administered every 3 months or less.
  Scores on the MoCA range from 0 to 30, with a score of 26 and higher generally considered normal. Population: Only measuring participants who completed the intervention. Measure is divided in two groups - 1) participants recruited pre-Covid 19 pandemic restrictions (maximum score of 30), and 2) Participants recruited after Covid 19 restrictions (maximum score of 22)
  units on a scale
    pre-Covid 19 restrictions: number analyzed (Participants) | 8
    pre-Covid 19 restrictions | 22.6 [10 to 27]
    post-Covid 19 restrictions: number analyzed (Participants) | 4
    post-Covid 19 restrictions | 17.75 [13 to 21]
Albert's Test [Count of Participants; unit: Participants] — Albert's Test is a screening tool used to detect the presence of unilateral spatial neglect (USN) in patients with stroke. In this test, patients must cross out lines that are placed in random orientations on a piece of paper. USN is indicated when lines are left uncrossed on the same side of the page as the patients motor deficit or brain lesion is located.
  Results are based on the number of lines left uncrossed on each side of the test sheet. If any lines are left uncrossed, and more than 70% of uncrossed lines are on the same side as motor deficit, USN is indicated. Population: Only measuring participants who completed the intervention.
  Participants
    number analyzed (Participants) | 12
    (all) | 2
Visual Analog Scale for Pain [Mean (Full Range); unit: units on a scale] — Ask patients to rate their arm pain on a scale of 0-10 (0 = no pain; 10 = unbearable pain) Population: Only measuring participants who completed the intervention.
  units on a scale
    number analyzed (Participants) | 12
    (all) | 0.8 [0 to 2.5]
EQ 5D 5L (Health related quality of life) [Mean (Full Range); unit: units on a scale] — Descriptive system using 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 possible values: 1 no problems, 2 slight problems, 3 moderate problems, 4 severe problems, and 5 extreme problems. Patient is asked to assign a value to each dimension. The digits for the 5 dimensions are combined into a 5-digit number describing the patient's health state. An index value is derived from the health state ranging from -0.285 (value of 5 on all dimensions) to 1 (value of 1 on all dimensions). Higher index values indicate better outcomes. Population: Only measuring participants who completed the intervention.
  units on a scale
    number analyzed (Participants) | 12
    (all) | 0.462 [-0.186 to 0.768]
mRankin [Mean (Full Range); unit: units on a scale] — Modified Rankin Scale for Neurologic Disability (mRankin) measures degree of disability in daily activities of people who have suffered a stroke. Scale ranges from 0-6, where 0=no symptoms at all; 1= No significant disability despite symptoms; 2=Slight disability; unable to do all previous activities, but able to look after own affairs unassisted; 3=Moderate disability; requiring some help, but able to walk unassisted; 4=Moderately severe disability; unable to walk and attend to bodily needs unassisted; 5=Severe disability; bedridden, incontinent and requiring constant nursing care; 6=Dead Population: Only measuring participants who completed the intervention.
  units on a scale
    number analyzed (Participants) | 12
    (all) | 2.8 [1 to 4]
Fugl-Meyer Assessment for upper extremity (FMA-UE) [Mean (Standard Deviation); unit: units on a scale] — The Fugl-Meyer Assessment for upper extremity (FMA-UE) has been tested extensively, and is found to have excellent psychometric properties. It is considered to assess the body function according to the International Classification of Functioning, Disability and Health (ICF).
  The FMA-UE is scored on a scale 0 - 66 points (a higher score indicates lower arm impairment) and is recommended as core measures to be used in every stroke recovery and rehabilitation trial. Population: Only measuring participants completing the intervention
  units on a scale
    number analyzed (Participants) | 12
    (all) | 37.7 (17.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Finding the OnTrack Intervention Acceptable in Semi Structured Interviews
Description: Semi structured interviews will involve gaining patients opinions on the strengths and weaknesses of OnTrack. Interviews determine whether participants found the intervention easy to use and acceptable and if it is fit for their rehabilitation needs.
Time Frame: Week 13
Population: Semi-structured interviews on participants who finished the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | OnTrack
Number analyzed (Participants) | 12
Participants | 12

2. Primary Outcome: Number of Therapists Finding the OnTrack Intervention Acceptable in Semi Structured Interviews
Description: To assess the feasibility of the study design and procedures. Semi structured interviews will aim to collect therapists opinions on the strengths and weaknesses of On-Track.
Time Frame: Week 13
Measure: Count of Participants; unit: Participants
Groups:
- Recruiting Therapists: Therapists responsible for identifying and recruiting participants to the study.
Arm/Group | Recruiting Therapists
Number analyzed (Participants) | 13
Participants | 6

3. Secondary Outcome: Modified Rankin Scale
Description: The modified Rankin Scale is the most prevalent functional outcome measure in contemporary stroke trials. The mRS quantifies disability using an ordinal hierarchical grading from 0 (no symptoms) to 5 (severe disability). A lower number indicates lower disability.
Time Frame: Baseline, follow-up (week 7), follow-up (week 13)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On-Track
Number analyzed (Participants) | 12
units on a scale
  Baseline | 2.8 (1.1)
  Follow-up 1 (week 7) | 2.5 (0.8)
  Follow-up 2 (week 13) | 1.9 (0.9)

4. Secondary Outcome: Fugl-Meyer Assessment for Upper Extremity (FMA-UE)
Description: The Fugl-Meyer Assessment for upper extremity (FMA-UE) has been tested extensively, and is found to have excellent psychometric properties. It is considered to assess the body function according to the International Classification of Functioning, Disability and Health (ICF).
  The FMA-UE is scored on a scale 0 - 66 points (a higher score indicates lower arm impairment) and is recommended as core measures to be used in every stroke recovery and rehabilitation trial.
Time Frame: Baseline, follow-up (week 7), follow-up (week 13)
Population: Collection of this outcome measure was suspended after the study went to a fully remote delivery method due to the outbreak of the Covid 19 pandemic. This outcome measure is not possible to administer remotely.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On-Track
Number analyzed (Participants) | 7
units on a scale
  Baseline | 37.7 (17.2)
  Follow up 1 (week 7) | 39 (20.1)
  Follow up 2 (week 13) | 36.4 (22.4)

5. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: The MoCA is a brief cognitive screening tool with high sensitivity and specificity for detecting mild cognitive impairment. The MoCA uses a 0-30 score scale and defines impairment as follows: score of 18-25=mild, 10-17=moderate and <10 = severe. A version of the test that can be applied remotely was used after the study went fully remote due to the Coronavirus pandemic; the remote version uses a 0-22 score and impairment as follows: 13-18=mild, 7-12=moderate, and <7 severe.
Time Frame: Baseline, follow-up (week 7), follow-up (week 13)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On-Track
Number analyzed (Participants) | 12
units on a scale
  Full test cohort - Baseline | 22.6 (6.9)
  Full test cohort - Follow up 1 (week 7) | 24 (5.1)
  Full test cohort - Follow up 2 (week 13) | 25.3 (1)
  Remote test cohort - Baseline | 17.8 (3.4)
  Remote test cohort - Follow up 1 (week 7) | 19 (1.9)
  Remote test cohort - Follow up 2 (week 13) | 18.3 (2.4)

6. Secondary Outcome: Unilateral Spatial Neglect (USN) (Aka Albert's Test)
Description: Albert's Test is a screening tool used to detect the presence of unilateral spatial neglect (USN) in patients with stroke. In this test, a series of 40 black lines, each about 2 cm long, are randomly oriented on a sheet of white A4 size paper in 6 rows. The test sheet is presented to the patient at their midline. The examiner asks the patient to cross out all of the lines, and demonstrates what is required by crossing out the 5 central lines. The patient is encouraged to cross out all the lines until satisfied that they have all been crossed.
  If any lines are left uncrossed, and more than 70% of uncrossed lines are on the same side as motor deficit, USN is indicated.
Time Frame: Baseline, follow-up (week 7), follow-up (week 13)
Measure: Count of Participants; unit: Participants
Arm/Group | On-Track
Number analyzed (Participants) | 12
Participants
  Baseline | 2
  Follow up 1 (week 7) | 1
  Follow up 2 (week 13) | 1

7. Secondary Outcome: System Usability Scale (SUS)
Description: The test is a simple, 10-item scale covering a variety of aspects of system usability, such as the need for support, training and complexity, and thus have a high level of face validity for measuring the usability of a system. The scale is from 0-100, a higher number signifies better usability.
Time Frame: Week 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | On-Track
Number analyzed (Participants) | 12
score on a scale | 84.6 (13.1)

8. Secondary Outcome: Patient Activation and Motivation (PAM) - Questionnaire 10 Short Questions
Description: The Patient Activation Measure (PAM) is a 10-item survey that assesses a person's underlying knowledge, skills and confidence integral to managing his or her own health and healthcare.
  PAM segments individuals into one of four activation levels along an empirically derived 100-point scale (0 min - 100 max, a higher score indicates a higher level of activation). Each level provides insight into an extensive array of health-related characteristics, including attitudes, motivators, and behaviors. Individuals in the lowest activation level do not yet understand the importance of their role in managing their own health, and have significant knowledge gaps and limited self-management skills. Individuals in the highest activation level are proactive with their health, have developed strong self- management skills, and are resilient in times of stress or change.
Time Frame: Baseline, follow-up (week 7), follow-up (week 13)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OnTrack
Number analyzed (Participants) | 12
units on a scale
  Baseline | 69.7 (17.8)
  Follow up 1 (week 7) | 65.8 (14.8)
  Follow up 2 (week 13) | 68.1 (10.3)

9. Secondary Outcome: Motor Assessment Log (MAL) - Questionnaire
Description: Structured interview intended to examine How Much and How Well the subject uses their more-affected arm outside of the laboratory setting. Standardized questions are asked about the amount of use of their more-affected arm (Amount Scale or AS) and the quality of their movement (How Well Scale or HW) during the functional activities. Two scales are printed on sheets of paper and are placed in front of the participant during test administration. Both scales range between 0 and 5 (half scores are possible, i.e. 0.5,1.5,2.5,3.5,4.5). Higher values represent a better outcome.
Time Frame: Baseline, follow-up (week 7), follow-up (week 13)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OnTrack
Number analyzed (Participants) | 12
score on a scale
  Baseline - How Well Scale | 2.26 (1.5)
  Baseline - Amount Scale | 2.00 (1.4)
  Follow up 1 (week 7) - How Well Scale | 3.09 (1.2)
  Follow up 1 (week 7) - Amount Scale | 2.94 (1.2)
  Follow up 2 (week 13) - How Well Scale | 3.17 (1.2)
  Follow up 2 (week 13) - Amount Scale | 3.24 (1.3)

10. Secondary Outcome: Visual Analogue Scale for Pain - Question
Description: Ask patients to rate their arm pain on a scale of 0-10 (0 = no pain; 10 = unbearable pain)
Time Frame: Baseline, follow-up (week 7), follow-up (week 13)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OnTrack
Number analyzed (Participants) | 12
score on a scale
  Baseline | 0.8 (1.0)
  Follow up 1 (week 7) | 2.5 (1.9)
  Follow up 2 (week 13) | 2.8 (2.3)

11. Secondary Outcome: Friends and Family Test
Description: Asks patient if they would recommend the service they have just received to friends/family. The NHS Friends and Family Test (FFT) was created to help service providers and commissioners understand whether patients are happy with the service provided, or where improvements are needed. 5 point Likert scale questionnaire ranging from 1-5: 1 "extremely unlikely", 2 "unlikely", 3 "neither likely nor unlikely", 4 "likely", 5 "extremely likely", an "I don't know" option is also provided. Higher values represent better outcomes.
Time Frame: Week 13
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | OnTrack
Number analyzed (Participants) | 12
score on a scale | 4.7 [4 to 5]

12. Secondary Outcome: EQ 5D 5L (Health Related Quality of Life)
Description: Descriptive system using 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 possible values: 1 no problems, 2 slight problems, 3 moderate problems, 4 severe problems, and 5 extreme problems. Patient is asked to assign a value to each dimension. The digits for the 5 dimensions are combined into a 5-digit number describing the patient's health state. An index value is derived from the health state ranging from -0.285 (value of 5 on all dimensions) to 1 (value of 1 on all dimensions). Higher index values indicate better outcomes.
Time Frame: Baseline, week 7, week 13
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | OnTrack
Number analyzed (Participants) | 12
score on a scale
  Baseline | 0.462 [-0.186 to 0.768]
  Follow-up 1 (week 7) | 0.585 [0.263 to 0.837]
  Follow-up 2 (week 13) | 0.606 [0.375 to 0.879]

ADVERSE EVENTS:
Time Frame: 20 months
Description: Participants in the trial were at zero risk for all-cause mortality and serious adverse events stemming from using the intervention or participating in the trail
Arm/Group | OnTrack
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT03944486/Prot_SAP_000.pdf